CLINICAL TRIAL: NCT00564876
Title: Phase II Study Evaluating The Safety And Response To Neoadjuvant Dasatinib In Early Stage Non-Small Cell Lung Cancer (NSCLC).
Brief Title: Phase II Study Evaluating The Safety And Response To Neoadjuvant Dasatinib In Early Stage Non-Small Cell Lung Cancer
Acronym: TOP0706
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual, study closed.
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001278
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non Small Cell Lung Cancer (NSCLC); carcinoma; dasatinib; neoadjuvant; adjuvant; resection; genomic signature; predictor; microarray
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Neoadjuvant dasatinib is to be administered as an oral dose of 70 mg PO twice daily on a continuous basis for 3 weeks prior to surgery. Patients will begin adjuvant dasatinib (70 mg PO twice daily) between 4-6 weeks after standard adjuvant therapy is complete or 4-8 weeks after surgery for those patients that do not receive adjuvant chemotherapy. Adjuvant dasatinib will be given on a continuous basis for up to 3 months after adjuvant chemotherapy or after surgery if no adjuvant chemotherapy is given.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Fresh frozen tumor tissue must be available prior to initiating dasatinib. Eligible patients will receive neoadjuvant dasatinib 70 mg PO twice daily for 3 weeks followed by surgery. The surgical specimen will be evaluated for pathologic response. The second tumor sample will be obtained after 3 weeks of dasatinib therapy at the time of definitive surgical resection which will be evaluated for changes in genomic expression profiles. Patients with at least a 15% decrease or better objective response, without evidence of progression (per tumor evaluation pre-surgery) or pathologic response (as defined as ≥30% tumor necrosis or cell death) to neoadjuvant dasatinib therapy will be eligible to receive dasatinib 70 mg twice daily for 90 days after the completion of standard adjuvant therapy.
  Other Names: Sprycel

SUMMARY:
Src expression has been identified in a majority of Non-Small Cell Lung Cancer (NSCLC) cell lines and there is preclinical evidence that Src family kinases may be important in hypoxic growth and angiogenesis in NSCLC. We hypothesize that the inhibition of Src pathway with dasatinib will demonstrate anti-tumor activity in early stage NSCLC, with a tolerable safety profile.

Patients will receive dasatinib, a Src inhibitor, for 3 weeks prior to surgical resection for early stage NSCLC. Fresh frozen tumor tissue is needed for genomic analysis. If fresh frozen tumor tissue is not available from the initial diagnosis, a biopsy will be required to participate in this trial. A second tumor sample will be obtained at time of surgical resection to evaluate for changes in genomic expression profiles.

Patients will be eligible to receive 3 months of adjuvant dasatinib therapy after completion of standard adjuvant therapy or after recovery from surgery if no standard adjuvant therapy is given, if there is evidence of neoadjuvant tumor response (radiologic and/or pathologic) to dasatinib.

Many patients who present with NSCLC are active smokers. Patients who are smoking up until the time of their surgery experience increased peri-operative complications compared to patients who have not smoked cigarettes immediately prior to surgery. While this trial will not be limited to active smokers, the period of smoking cessation prior to surgery is an attractive window of opportunity during which the potentially active novel anticancer therapy dasatinib can be offered to the patient.

DETAILED DESCRIPTION:
This is a phase II study of dasatinib, a targeted biologic agent, known to inhibit Src. It is difficult to assess outcome in phase II adjuvant trials because there is no measurable disease to evaluate efficacy and there are many variables that could confound comparing survival of subjects on trial to historical controls. Therefore, after a fresh frozen tumor tissue sample is obtained for genomic analysis, we plan to treat subjects with neoadjuvant dasatinib and then measure tumor response to therapy prior to surgery. Resected tumor will also be assessed for pathologic response as well as for changes in genomic expression patterns.

Subjects will be treated with neoadjuvant dasatinib 70 mg PO twice daily for 3 weeks, with a mandatory minimum of 3 days (72 hours) off of study drug prior to surgical resection. Imaging studies will be done pre-treatment and pre-surgery to assess radiologic response to therapy. The surgical specimen will be evaluated for pathologic response. A tumor tissue sample will be obtained from the surgical specimen for genomic analysis and will be evaluated for changes in genomic expression profiles.

Patients whose tumors have a response to neoadjuvant dasatinib therapy might benefit with better cancer control if they receive a potentially therapeutic course of adjuvant dasatinib. Patients that have at least a 15% decrease or better objective response, without evidence of progression to neoadjuvant dasatinib (per tumor evaluation pre-surgery) or pathologic response (as defined as ≥30% tumor necrosis or cell death) to neoadjuvant dasatinib therapy will be eligible to receive dasatinib 70 mg twice daily for 90 days after the completion of standard adjuvant therapy or after recovery from surgery if no standard adjuvant therapy is given. Patients will be followed for approximately 30 days after the last dose of dasatinib to assess toxicity.

Response will be evaluated in Src regulated and Src deregulated cohorts of tumors. If responses to neoadjuvant dasatinib occur, then accrual to either or both cohorts will be expanded. If there are no responses to neoadjuvant dasatinib in the cohort groups, then accrual to either or both cohorts will be stopped. The results of this study may be useful in designing future studies in early stage NSCLC using dasatinib alone or in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or histological/cytological diagnosis of Non-Small Cell Lung Cancer (NSCLC), Stage IB (≥4 cm per CT) or Stage IIA or IIB, amenable to surgical resection
* Must be deemed a surgical candidate
* Tumors ≥2 cm in maximum diameter without radiographic, bronchoscopic or pathologic evidence of nodal metastases are eligible for biopsy
* Fresh tissue biopsy material must be available for genomics analysis prior to initiating dasatinib therapy
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* No prior chemotherapy, immunotherapy, radiation therapy or biologic/targeted therapy for any malignancy
* Adequate Organ Function:

  * Total bilirubin <institutional upper limit normal (ULN)
  * Hepatic enzymes (AST, ALT) ≤2.5x institutional ULN
  * Serum creatinine <1.5x institutional ULN
  * Hemoglobin ≥9 gm/dL
  * Neutrophil count (ANC or AGC) ≥1500 per μL
  * Platelets ≥100,000 per μL
  * Prothrombin time (PT)/a partial thromboplastin time (PTT) ≤1.5x control
* No other serious medical or psychiatric illness
* Ability to take oral medication (dasatinib must be swallowed whole)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test preferably within 72 hours and no later than 7 days, prior to the start of study drug administration
* Both sexually active males and females of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped
* Signed written informed consent including Health Insurance Portability and Accountability Act (HIPAA) according to institutional guidelines

Exclusion Criteria:

* Previous or concomitant malignancy in the past 2 years other than curatively treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin
* Prior dasatinib therapy
* Evidence of pleural or pericardial effusion of any grade
* Cardiac Symptoms:

  * Uncontrolled angina, congestive heart failure (CHF), or myocardial infarction (MI) within 6 months
  * Diagnosed congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes)
  * Prolonged QT corrected (QTc) interval on pre-entry EKG (>450 msec)
  * Uncontrolled hypertension defined as >160/90 on a regimen of antihypertensive therapy
* Subjects with hypokalemia or hypomagnesaemia if it cannot be corrected
* History of diagnosed congenital acquired bleeding disorders (e.g., von Willebrand's disease)
* Ongoing or recent (≤3 months) significant (≥grade 3) gastrointestinal bleeding
* Concomitant Medications:

  * Drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)

    **quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
  * Current therapeutic dose heparin or coumadin therapy
  * St. John's Wort and all herbal supplements must be stopped while on dasatinib
  * IV bisphosphonates will be withheld for 2 weeks prior and 6 weeks after dasatinib administration due to risk of hypocalcaemia
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
* Pregnant or breastfeeding
* Active or uncontrolled infection requiring intravenous antibiotics
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dasatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patients who have received investigational drugs ≤4 weeks prior to starting study drug and/or who have not recovered from side effects of such therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Genomic signatures to guide the use of chemotherapeutics. Nat Med. 2006 Nov;12(11):1294-300. doi: 10.1038/nm1491. Epub 2006 Oct 22. PMID 17057710 (Retraction: PMID 21217686 Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Nat Med. 2011 Jan;17(1):135)
- [Background] Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. A genomic strategy to refine prognosis in early-stage non-small-cell lung cancer. N Engl J Med. 2006 Aug 10;355(6):570-80. doi: 10.1056/NEJMoa060467. PMID 16899777 (Retraction: PMID 21366430 Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. N Engl J Med. 2011 Mar 24;364(12):1176)
- [Background] Huang E, Ishida S, Pittman J, Dressman H, Bild A, Kloos M, D'Amico M, Pestell RG, West M, Nevins JR. Gene expression phenotypic models that predict the activity of oncogenic pathways. Nat Genet. 2003 Jun;34(2):226-30. doi: 10.1038/ng1167. PMID 12754511
- See also: Clinical Trials at Duke Comprehensive Cancer Center — http://www.cancer.duke.edu/CTrials/index.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to poor enrollment, this trial was closed to accrual and thus no results came from this trial.
Groups:
- Neoadjuvant Dasatinib: Neoadjuvant dasatinib is to be administered as an oral dose of 70 mg PO twice daily on a continuous basis for 3 weeks prior to surgery. Patients will begin adjuvant dasatinib (70 mg PO twice daily) between 4-6 weeks after standard adjuvant therapy is complete or 4-8 weeks after surgery for those patients that do not receive adjuvant chemotherapy. Adjuvant dasatinib will be given on a continuous basis for up to 3 months after adjuvant chemotherapy or after surgery if no adjuvant chemotherapy is given.
Period: Overall Study
Arm/Group | Neoadjuvant Dasatinib
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Dasatinib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2
Dasatinib [Number; unit: participants] — 70 mg dasatinib orally twice daily for 3 weeks
  participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate (radiologic and pathologic) in Stage IB and II to neoadjuvant dasatinib
Time Frame: First progression and survival every 3 months for 2 years, then every 6 months until 5 years, then yearly.
Arm/Group | Neoadjuvant Dasatinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety and Tolerability of Neoadjuvant Dasatinib
Description: Determine the safety and tolerability of neoadjuvant dasatinib in early stage NSCLC.
Time Frame: Screening / Baseline; Neoadjuvant dasatinib Cycle 1 Day 1 and Day 22
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Neoadjuvant Dasatinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Gene Expression Profile Activation of Src Pathways
Description: Determine whether gene expression profile activation of Src pathways is correlated with anti-tumor activity of dasatinib in early stage NSCLC.
Time Frame: Baseline and after 3 weeks of dasatinib therapy at the time of definitive surgical resection.
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Neoadjuvant Dasatinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Tolerability of Adjuvant Dasatinib
Description: Determine the safety and tolerability of adjuvant dasatinib in early stage NSCLC.
Time Frame: Duration of adjuvant treatment plus 30 days.
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Neoadjuvant Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Neoadjuvant Dasatinib
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Limitations for this trial were the trial was stopped due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No